CLINICAL TRIAL: NCT02584153
Title: An Open-label, Single-arm, Phase 1 Study Examining the Safety and Efficacy of Fibrin Sealant Plus Silver Microparticles to Prevent Incisional Hernias (HiP_1 Trial) Following Abdominal Surgery
Brief Title: A Study of Fibrin Sealant Plus Silver Microparticles to Prevent Incisional Hernias Following Abdominal Surgery
Acronym: HiP_1
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Did not obtain IND or IRB approval to initiate study.
Sponsor: Hobart Harris (Other)
Responsible Party: Sponsor-Investigator, Hobart Harris, Professor & Chief, Division of General Surgery, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HiP_1
Record Dates: First submitted 2015-10-19; First posted 2015-10-22 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Hernia; Ventral Hernia; Abdominal Hernia
Keywords: Hernia; Ventral; Incisional; Abdominal; Herniorrhaphy; Recurrence; laparotomy; prevention
MeSH Terms: conditions — Hernia; Hernia, Ventral; Hernia, Abdominal; Surgical Wound; Recurrence | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Myoseal (Experimental): The fibrin sealant and silver microparticles are sprayed onto the surface of the sutured myofascial incision following abdominal surgery.
  Interventions: Drug: Fibrin Sealant; Drug: Silver Microparticles

INTERVENTIONS:
Drug: Fibrin Sealant — TISSEEL® fibrin sealant (Baxter Biosurgery, Deerfield, IL)
  Other Names: TISSUCOL/TISSEEL STIM3; TISSUCOL/TISSEEL STIM4; Fibrin Sealant VH S/D
Drug: Silver Microparticles — Product Code: AG-M-04M-P.200M (American Elements, Los Angeles, CA)
  Other Names: Ag

SUMMARY:
Incisional hernias are a frequent consequence of abdominal surgery. Current clinical efforts are primarily focused on improving repair materials and surgical techniques to correct these hernias instead of the optimal solution: prevention.

A product called MYOSEAL is currently being developed to prevent hernia formation after abdominal surgery by using fibrin tissue sealant and silver particles to prophylactically enhance the early wound healing of myofascial incisions. The purpose of this phase 1 study is to examine the safety of applying MYOSEAL immediately after abdominal wall suture closure in patients undergoing abdominal surgery. The investigators expect that applying this product to sutured myofascial incisions will increase collagen formation in the wound and thus prevent the formation of incisional hernias.

DETAILED DESCRIPTION:
Hernias are areas of weakness in the muscle of the abdomen and commonly develop after people have had abdominal surgery. This area of weakness often turns into a bulge or protrusion that can increase in size over time, interfere with the intestines and make it difficult for people to work or exercise. Many people undergo surgery to fix their hernia. Unfortunately, the operations to repair the hernia frequently fail and the hernia returns. The investigators are developing a material to help the body heal after abdominal surgery and thereby prevent incisional hernias for forming in the first place. This study is the first step in testing this new material in patients and whether it is safe to use. This study will include patients having all types of abdominal surgeries.

The test material is called MYOSEAL; a combination of a tissue sealant called TISSEEL® (Baxter Biosurgery, Deerfield, IL) plus small particles of metallic silver (<250µ, American Elements, Los Angeles, CA). TISSEEL is made from naturally occurring blood proteins and has been approved by the Food and Drug Administration (FDA) for use in surgery since 1998. But, TISSEEL has not been approved to prevent incisional hernias after abdominal surgery. The silver particles are not approved by FDA, but are thought to be generally safe in the way they will be used. This study hopes to learn how to help the body better heal after abdominal surgery.

At the conclusion of a laparotomy, 4-6 pairs of stainless steel clips (large Horizon® titanium clips, Teleflex Medical, Research Triangle Park, NC) will be attached opposite each other and equally spaced to the edges of the sutured myofascial incision, followed by the application of MYOSEAL to the sutured myofascial incision before closure of the skin. Study participants will be examined at 1 day, 1 month, 3 months, and 6 months after surgery. The primary endpoints include wound occurrences, including wound infections, seromas, and hematomas and postoperative complications through 6 months following surgery. The secondary endpoint is the incisional hernia rate at 1 month as determined by the distance between the metal clips marking the myofascial edges using calipers and a plain abdominal radiograph.

ELIGIBILITY:
Inclusion Criteria:

* The patient is undergoing an abdominal operation requiring an incision ≥10-cm in length;
* Age ≥21;
* Negative pregnancy test;
* No allergic, religious or ethical objections to fibrin tissue sealants (human blood proteins), aprotinin or metallic silver;
* Signed informed consent to take part in the study

Exclusion Criteria:

* Lactating women;
* Patients who are unable to commit to the follow evaluations over 6 months;
* Severe malnutrition (serum albumin <2.0);
* Use of an investigational agent within 1 month prior to study enrollment and/or planned during this study;
* Immunocompromised patients, as evidenced by: administration of high doses of corticosteroids (i.e. doses ≥ 1.5 mg/kg/day of prednisone or equivalent) within 72 hours before study enrollment; status post solid organ transplant or bone marrow transplant AND experiencing acute organ rejection or bone marrow failure or rejection; evidence of neutropenia (absolute neutrophil count ≤ 500 cells/mm3 (≤ 500 x 106 cells/L); immunosuppression secondary to immunomodulatory medications (e.g. cyclosporin, azathioprine, OKT3), chemotherapy or radiation therapy within 90 days before study enrollment; known AIDS; any disease sufficiently advanced to suppress resistance to infection (including, but not limited to leukemia, lymphoma or hypogammaglobulinemia); administration of immunoglobulin of G-CSF within 90 days before study enrollment;
* Presence of an underlying disease/injury with life expectancy less than two years and/or severe underlying disease that would preclude study entry (e.g. known malignancy).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Wound Occurrences | 6 months after surgery
  Wound events include surgical site infections as well as seromas/hematomas.
Post-operative Complications | 6 months after surgery
  Post-operative complications include urinary tract infection and sepsis.

SECONDARY OUTCOMES:
Incisional Hernia | 1 month after surgery
  Incisional hernia as determined by the distance between the metal clips marking the myofascial edges on abdominal radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Hobart W. Harris, M.D., M.P.H., Principal Investigator — University of California, San Francisco